CLINICAL TRIAL: NCT05601856
Title: Gut Microbiome and Blood Indices in Patients With AD and Their Spousal Caregivers
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Zhiyi Zuo, MD, Professor, Anesthesiology, University of Virginia
Other Study IDs: HSR220333
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; Gut Biome
Keywords: Alzheimers; biome
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Serum, 5 mL Stool Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Alzheimer's Patient: patients with AD whose clinical dementia rating (CDR) is > 1 Age 65-90 with none of the criteria below:
  1. Familial Alzheimer's Disease (AD)
  2. Severe cardiovascular disease
  3. Severe respiratory system disease
  4. Severe liver disease
  5. Severe kidney disease
  6. Severe central nervous system diseases
  7. Having a lifespan of fewer than 3 months
  8. History of psychiatric illness
  9. Major neurological diseases other than AD
  10. Current use of corticosteroids, antibiotics, or bowel motility modification agents
  11. Any history of Alcoholism or illicit drug dependence
  12. Previous inclusion in this study
  13. Difficulty with follow-up or poor compliance
  14. Severe hearing impairment
  15. Severe vision impairment
- Spousal Caregiver to Alzheimer's Patient: Spousal Caregiver to "Alzheimer's Patient" group, Age 65-90 with none of the criteria below:
  1. Familial Alzheimer's Disease (AD)
  2. Severe cardiovascular disease
  3. Severe respiratory system disease
  4. Severe liver disease
  5. Severe kidney disease
  6. Severe central nervous system diseases
  7. Having a lifespan of fewer than 3 months
  8. History of psychiatric illness
  9. Major neurological diseases other than AD
  10. Current use of corticosteroids, antibiotics, or bowel motility modification agents
  11. Any history of Alcoholism or illicit drug dependence
  12. Previous inclusion in this study
  13. Difficulty with follow-up or poor compliance
  14. Severe hearing impairment
  15. Severe vision impairment
- Healthy adult control: Age-matched to "Spousal Caregiver to Alzheimer's Patient" group Age 65-90 with none of the criteria below:
  1. Familial Alzheimer's Disease (AD)
  2. Severe cardiovascular disease
  3. Severe respiratory system disease
  4. Severe liver disease
  5. Severe kidney disease
  6. Severe central nervous system diseases
  7. Having a lifespan of fewer than 3 months
  8. History of psychiatric illness
  9. Major neurological diseases other than AD
  10. Current use of corticosteroids, antibiotics, or bowel motility modification agents
  11. Any history of Alcoholism or illicit drug dependence
  12. Previous inclusion in this study
  13. Difficulty with follow-up or poor compliance
  14. Severe hearing impairment
  15. Severe vision impairment

SUMMARY:
Spousal caregivers of Alzheimer's Dementia (AD) patients have an elevated risk of developing AD in the future. Past studies have shown the presence of serum indicators correlated with gut biome dysfunction in AD patients. We hypothesize that the same gut biome dysfunction may be present in spousal caregivers of AD patients.

DETAILED DESCRIPTION:
Patients with Alzheimer's disease (AD) have gut dysbiosis. Short-chain fatty acids (SCFAs) are products of the gut microbiome. Among them, Acetate and valeric acid were positively correlated with the Aβ plaque load detected by amyloid PET in participants with or without AD. However, the levels of SCFAs in the blood of patients with AD have not been defined. Also, the usefulness of indices of inflammation and neuropathology in the blood as biomarkers for cognitive impairment in patients with AD is elusive. Importantly, spousal caregivers of patients with dementia have a higher risk of developing dementia later in life than those whose spouses do not have dementia. The spousal caregivers have an accelerated cognitive decline. The mechanisms for these phenomena are not known. We hypothesize that spousal caregivers of patients with AD have gut microbiome and levels of blood SCFAs similar to those of patients with AD, that these spouses have increased inflammatory cytokines and indices of AD-like neuropathology in the blood, and that there is a correlation between the cognition and various indices in the blood among patients with AD, their spouses, and age-matched controls. To address these hypotheses, we will recruit three groups of participants: Patients with AD, their spousal caregivers, and controls that are age-matched with the caregivers. Their gut microbiome and indices of neuroinflammation and neuropathology in the blood will be determined. Their cognition will be assessed. The correction of cognition with gut microbiome genera or indices in the blood will be analyzed. Our studies may represent the first study to determine whether the gut microbiome and SCFAs may play a role in the cognitive impairment in the spousal caregivers of patients with AD. These studies may also identify biomarkers for cognitive impairment in these caregivers and patients with AD. These findings may ultimately help the care of patients with AD and reduce the cognitive declines in spousal caregivers of patients with AD.

ELIGIBILITY:
Inclusion Criteria:

1. patients with AD whose clinical dementia rating (CDR) is > 1
2. Spouses of Patients in the above group Or
3. Healthy adult unrelated to groups 1 and 2, with no history of dementia And
4. Regardless of the grouping, the prospective subject must be between 65 and 90 years old

Exclusion Criteria:

1. Familial Alzheimer's Disease (AD)
2. Severe cardiovascular disease
3. Severe respiratory system disease
4. Severe liver disease
5. Severe kidney disease
6. Severe central nervous system diseases
7. Having a lifespan of fewer than 3 months
8. History of psychiatric illness
9. Major neurological diseases other than AD
10. Current use of corticosteroids, antibiotics, or bowel motility modification agents
11. Any history of Alcoholism or illicit drug dependence
12. Previous inclusion in this study
13. Difficulty with follow-up or poor compliance
14. Severe hearing impairment
15. Severe vision impairment

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults who are at risk for Alzheimer's Disease.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Inflammation related biomarkers | one day
  interleukin (IL)-1β, IL-6, IL-10, IL-17, complement 3 (C3,) and YKL-40
amyloid biomarker | one day
  amyloid beta (Aβ)1-42
ratio of Aβ1-42 and Aβ1-40 | one day
total tau biomarker | one day
phospho-tau at 181 or 217 biomarker | one day
neurodegeneration related biomarkers | one day
  neurofilament light chain (NFL) and neurogranin
serum short chain fatty acids | one day
  acetic acid, propionic acid, isobutyric acid, butyric acid, valeric acid and hexanic acid

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
If shared, it will be de-identified data.

REFERENCES:
- [Background] Vassar R, Citron M. Abeta-generating enzymes: recent advances in beta- and gamma-secretase research. Neuron. 2000 Sep;27(3):419-22. doi: 10.1016/s0896-6273(00)00051-9. No abstract available. PMID 11055423
- [Background] Vassar R. BACE1: the beta-secretase enzyme in Alzheimer's disease. J Mol Neurosci. 2004;23(1-2):105-14. doi: 10.1385/JMN:23:1-2:105. PMID 15126696
- [Background] Selkoe DJ. Alzheimer's disease: genes, proteins, and therapy. Physiol Rev. 2001 Apr;81(2):741-66. doi: 10.1152/physrev.2001.81.2.741. PMID 11274343
- [Background] Wang WY, Tan MS, Yu JT, Tan L. Role of pro-inflammatory cytokines released from microglia in Alzheimer's disease. Ann Transl Med. 2015 Jun;3(10):136. doi: 10.3978/j.issn.2305-5839.2015.03.49. PMID 26207229
- [Background] Saji N, Murotani K, Hisada T, Tsuduki T, Sugimoto T, Kimura A, Niida S, Toba K, Sakurai T. The relationship between the gut microbiome and mild cognitive impairment in patients without dementia: a cross-sectional study conducted in Japan. Sci Rep. 2019 Dec 18;9(1):19227. doi: 10.1038/s41598-019-55851-y. PMID 31852995
- [Background] Guo M, Peng J, Huang X, Xiao L, Huang F, Zuo Z. Gut Microbiome Features of Chinese Patients Newly Diagnosed with Alzheimer's Disease or Mild Cognitive Impairment. J Alzheimers Dis. 2021;80(1):299-310. doi: 10.3233/JAD-201040. PMID 33523001
- [Background] Wang X, Sun G, Feng T, Zhang J, Huang X, Wang T, Xie Z, Chu X, Yang J, Wang H, Chang S, Gong Y, Ruan L, Zhang G, Yan S, Lian W, Du C, Yang D, Zhang Q, Lin F, Liu J, Zhang H, Ge C, Xiao S, Ding J, Geng M. Sodium oligomannate therapeutically remodels gut microbiota and suppresses gut bacterial amino acids-shaped neuroinflammation to inhibit Alzheimer's disease progression. Cell Res. 2019 Oct;29(10):787-803. doi: 10.1038/s41422-019-0216-x. Epub 2019 Sep 6. PMID 31488882
- [Background] Kim MS, Kim Y, Choi H, Kim W, Park S, Lee D, Kim DK, Kim HJ, Choi H, Hyun DW, Lee JY, Choi EY, Lee DS, Bae JW, Mook-Jung I. Transfer of a healthy microbiota reduces amyloid and tau pathology in an Alzheimer's disease animal model. Gut. 2020 Feb;69(2):283-294. doi: 10.1136/gutjnl-2018-317431. Epub 2019 Aug 30. PMID 31471351
- [Background] Li B, He Y, Ma J, Huang P, Du J, Cao L, Wang Y, Xiao Q, Tang H, Chen S. Mild cognitive impairment has similar alterations as Alzheimer's disease in gut microbiota. Alzheimers Dement. 2019 Oct;15(10):1357-1366. doi: 10.1016/j.jalz.2019.07.002. Epub 2019 Aug 18. PMID 31434623
- [Background] Lai Z, Shan W, Li J, Min J, Zeng X, Zuo Z. Appropriate exercise level attenuates gut dysbiosis and valeric acid increase to improve neuroplasticity and cognitive function after surgery in mice. Mol Psychiatry. 2021 Dec;26(12):7167-7187. doi: 10.1038/s41380-021-01291-y. Epub 2021 Oct 18. PMID 34663905
- [Background] Liu H, McPherson BC, Zhu X, Da Costa ML, Jeevanandam V, Yao Z. Role of nitric oxide and protein kinase C in ACh-induced cardioprotection. Am J Physiol Heart Circ Physiol. 2001 Jul;281(1):H191-7. doi: 10.1152/ajpheart.2001.281.1.H191. PMID 11406485
- [Background] Colombo AV, Sadler RK, Llovera G, Singh V, Roth S, Heindl S, Sebastian Monasor L, Verhoeven A, Peters F, Parhizkar S, Kamp F, Gomez de Aguero M, MacPherson AJ, Winkler E, Herms J, Benakis C, Dichgans M, Steiner H, Giera M, Haass C, Tahirovic S, Liesz A. Microbiota-derived short chain fatty acids modulate microglia and promote Abeta plaque deposition. Elife. 2021 Apr 13;10:e59826. doi: 10.7554/eLife.59826. PMID 33845942
- [Background] Marizzoni M, Cattaneo A, Mirabelli P, Festari C, Lopizzo N, Nicolosi V, Mombelli E, Mazzelli M, Luongo D, Naviglio D, Coppola L, Salvatore M, Frisoni GB. Short-Chain Fatty Acids and Lipopolysaccharide as Mediators Between Gut Dysbiosis and Amyloid Pathology in Alzheimer's Disease. J Alzheimers Dis. 2020;78(2):683-697. doi: 10.3233/JAD-200306. PMID 33074224
- [Background] Norton MC, Smith KR, Ostbye T, Tschanz JT, Corcoran C, Schwartz S, Piercy KW, Rabins PV, Steffens DC, Skoog I, Breitner JC, Welsh-Bohmer KA; Cache County Investigators. Greater risk of dementia when spouse has dementia? The Cache County study. J Am Geriatr Soc. 2010 May;58(5):895-900. doi: 10.1111/j.1532-5415.2010.02806.x. PMID 20722820
- [Background] Vitaliano PP, Zhang J, Scanlan JM. Is caregiving hazardous to one's physical health? A meta-analysis. Psychol Bull. 2003 Nov;129(6):946-72. doi: 10.1037/0033-2909.129.6.946. PMID 14599289
- [Background] Drouet B, Pincon-Raymond M, Chambaz J, Pillot T. Molecular basis of Alzheimer's disease. Cell Mol Life Sci. 2000 May;57(5):705-15. doi: 10.1007/s000180050035. PMID 10892337
- [Background] Gotz J, Streffer JR, David D, Schild A, Hoerndli F, Pennanen L, Kurosinski P, Chen F. Transgenic animal models of Alzheimer's disease and related disorders: histopathology, behavior and therapy. Mol Psychiatry. 2004 Jul;9(7):664-83. doi: 10.1038/sj.mp.4001508. PMID 15052274
- [Background] Heppner FL, Ransohoff RM, Becher B. Immune attack: the role of inflammation in Alzheimer disease. Nat Rev Neurosci. 2015 Jun;16(6):358-72. doi: 10.1038/nrn3880. PMID 25991443
- [Background] Dassel KB, Carr DC, Vitaliano P. Does Caring for a Spouse With Dementia Accelerate Cognitive Decline? Findings From the Health and Retirement Study. Gerontologist. 2017 Apr 1;57(2):319-328. doi: 10.1093/geront/gnv148. PMID 26582383
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Feldman HH, Frisoni GB, Hampel H, Jagust WJ, Johnson KA, Knopman DS, Petersen RC, Scheltens P, Sperling RA, Dubois B. A/T/N: An unbiased descriptive classification scheme for Alzheimer disease biomarkers. Neurology. 2016 Aug 2;87(5):539-47. doi: 10.1212/WNL.0000000000002923. Epub 2016 Jul 1. PMID 27371494
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Blennow K, Zetterberg H. Biomarkers for Alzheimer's disease: current status and prospects for the future. J Intern Med. 2018 Dec;284(6):643-663. doi: 10.1111/joim.12816. Epub 2018 Aug 19. PMID 30051512
- [Background] Hellwig K, Kvartsberg H, Portelius E, Andreasson U, Oberstein TJ, Lewczuk P, Blennow K, Kornhuber J, Maler JM, Zetterberg H, Spitzer P. Neurogranin and YKL-40: independent markers of synaptic degeneration and neuroinflammation in Alzheimer's disease. Alzheimers Res Ther. 2015 Dec 24;7:74. doi: 10.1186/s13195-015-0161-y. PMID 26698298
- [Background] Sharma N, Singh AN. Exploring Biomarkers for Alzheimer's Disease. J Clin Diagn Res. 2016 Jul;10(7):KE01-6. doi: 10.7860/JCDR/2016/18828.8166. Epub 2016 Jul 1. PMID 27630867
- [Background] Minter MR, Zhang C, Leone V, Ringus DL, Zhang X, Oyler-Castrillo P, Musch MW, Liao F, Ward JF, Holtzman DM, Chang EB, Tanzi RE, Sisodia SS. Antibiotic-induced perturbations in gut microbial diversity influences neuro-inflammation and amyloidosis in a murine model of Alzheimer's disease. Sci Rep. 2016 Jul 21;6:30028. doi: 10.1038/srep30028. PMID 27443609
- [Background] Bonfili L, Cecarini V, Berardi S, Scarpona S, Suchodolski JS, Nasuti C, Fiorini D, Boarelli MC, Rossi G, Eleuteri AM. Microbiota modulation counteracts Alzheimer's disease progression influencing neuronal proteolysis and gut hormones plasma levels. Sci Rep. 2017 May 25;7(1):2426. doi: 10.1038/s41598-017-02587-2. PMID 28546539
- [Background] Harach T, Marungruang N, Duthilleul N, Cheatham V, Mc Coy KD, Frisoni G, Neher JJ, Fak F, Jucker M, Lasser T, Bolmont T. Reduction of Abeta amyloid pathology in APPPS1 transgenic mice in the absence of gut microbiota. Sci Rep. 2017 Feb 8;7:41802. doi: 10.1038/srep41802. PMID 28176819
- [Background] Biagi E, Nylund L, Candela M, Ostan R, Bucci L, Pini E, Nikkila J, Monti D, Satokari R, Franceschi C, Brigidi P, De Vos W. Through ageing, and beyond: gut microbiota and inflammatory status in seniors and centenarians. PLoS One. 2010 May 17;5(5):e10667. doi: 10.1371/journal.pone.0010667. PMID 20498852
- [Background] Chen H, Meng L, Shen L. Multiple roles of short-chain fatty acids in Alzheimer disease. Nutrition. 2022 Jan;93:111499. doi: 10.1016/j.nut.2021.111499. Epub 2021 Sep 23. PMID 34735921
- [Background] Liu J, Li H, Gong T, Chen W, Mao S, Kong Y, Yu J, Sun J. Anti-neuroinflammatory Effect of Short-Chain Fatty Acid Acetate against Alzheimer's Disease via Upregulating GPR41 and Inhibiting ERK/JNK/NF-kappaB. J Agric Food Chem. 2020 Jul 8;68(27):7152-7161. doi: 10.1021/acs.jafc.0c02807. Epub 2020 Jun 25. PMID 32583667
- [Background] Killingsworth J, Sawmiller D, Shytle RD. Propionate and Alzheimer's Disease. Front Aging Neurosci. 2021 Jan 11;12:580001. doi: 10.3389/fnagi.2020.580001. eCollection 2020. PMID 33505301
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Sherwin E, Dinan TG, Cryan JF. Recent developments in understanding the role of the gut microbiota in brain health and disease. Ann N Y Acad Sci. 2018 May;1420(1):5-25. doi: 10.1111/nyas.13416. Epub 2017 Aug 2. PMID 28768369
- [Background] Olsson B, Lautner R, Andreasson U, Ohrfelt A, Portelius E, Bjerke M, Holtta M, Rosen C, Olsson C, Strobel G, Wu E, Dakin K, Petzold M, Blennow K, Zetterberg H. CSF and blood biomarkers for the diagnosis of Alzheimer's disease: a systematic review and meta-analysis. Lancet Neurol. 2016 Jun;15(7):673-684. doi: 10.1016/S1474-4422(16)00070-3. Epub 2016 Apr 8. PMID 27068280
- [Background] Cao L, Li L, Lin D, Zuo Z. Isoflurane induces learning impairment that is mediated by interleukin 1beta in rodents. PLoS One. 2012;7(12):e51431. doi: 10.1371/journal.pone.0051431. Epub 2012 Dec 12. PMID 23251531
- [Background] Wang Z, Meng S, Cao L, Chen Y, Zuo Z, Peng S. Critical role of NLRP3-caspase-1 pathway in age-dependent isoflurane-induced microglial inflammatory response and cognitive impairment. J Neuroinflammation. 2018 Apr 17;15(1):109. doi: 10.1186/s12974-018-1137-1. PMID 29665808
- [Background] Zhang J, Tan H, Jiang W, Zuo Z. Amantadine alleviates postoperative cognitive dysfunction possibly by increasing glial cell line-derived neurotrophic factor in rats. Anesthesiology. 2014 Oct;121(4):773-85. doi: 10.1097/ALN.0000000000000352. PMID 25251457
- [Background] Li H, Yin J, Li L, Deng J, Feng C, Zuo Z. Isoflurane postconditioning reduces ischemia-induced nuclear factor-kappaB activation and interleukin 1beta production to provide neuroprotection in rats and mice. Neurobiol Dis. 2013 Jun;54:216-24. doi: 10.1016/j.nbd.2012.12.014. Epub 2013 Jan 8. PMID 23313315
- [Background] Li J, Sheng W, Feng C, Zuo Z. Pyrrolidine dithiocarbamate attenuates brain Abeta increase and improves long-term neurological outcome in rats after transient focal brain ischemia. Neurobiol Dis. 2012 Jan;45(1):564-72. doi: 10.1016/j.nbd.2011.09.013. Epub 2011 Sep 24. PMID 21983158
- [Background] Watt G, Shang K, Zieba J, Olaya J, Li H, Garner B, Karl T. Chronic Treatment with 50 mg/kg Cannabidiol Improves Cognition and Moderately Reduces Abeta40 Levels in 12-Month-Old Male AbetaPPswe/PS1DeltaE9 Transgenic Mice. J Alzheimers Dis. 2020;74(3):937-950. doi: 10.3233/JAD-191242. PMID 32116258
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] Li Y, Chen D, Wang H, Wang Z, Song F, Li H, Ling L, Shen Z, Hu C, Peng J, Li W, Xing W, Pan J, Liang H, Zhou Q, Cai J, He Z, Peng S, Zeng W, Zuo Z. Intravenous versus Volatile Anesthetic Effects on Postoperative Cognition in Elderly Patients Undergoing Laparoscopic Abdominal Surgery. Anesthesiology. 2021 Mar 1;134(3):381-394. doi: 10.1097/ALN.0000000000003680. PMID 33439974